CLINICAL TRIAL: NCT04504149
Title: Patient Readiness for Improvement Through Motivation, Engagement, and Decision-making for PTSD (CDA 18-186)
Brief Title: Shared Decision Making for PTSD in Primary Care
Acronym: PRIMED-PTSD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Findings from Aims 1 and 2 clarified that any future trial should involve provider- or clinic-level randomization, not patient-level randomization.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CDX 20-002
Record Dates: First submitted 2020-07-29; First posted 2020-08-07 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: PTSD
Keywords: Primary Care; Decision Making, Shared; Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Patient Readiness for Improvement through Motivation, Engagement, and Decision-making for PTSD, hereafter PRIMED, is a primary care-based shared decision making (SDM) intervention that the investigators will develop using UCD methods for VA Primary Care-Mental Health Integration (PC-MHI) clinics to engage Veterans in first-line treatments for PTSD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRIMED (Experimental): Shared decision making session
  Interventions: Behavioral: Patient Readiness for Improvement through Motivation, Engagement, and Decision-making for PTSD
- Usual Care (No Intervention): The investigators will characterize usual care using chart review and administrative data to identify medications (prescribed, filled), number of mental health sessions received, types of providers seen, and the content of treatment sessions as captured in chart notes.

INTERVENTIONS:
Behavioral: Patient Readiness for Improvement through Motivation, Engagement, and Decision-making for PTSD — A primary care-based shared decision making intervention
  Other Names: PRIMED
  Arms: PRIMED

SUMMARY:
PTSD is one of the most common mental health conditions affecting Veterans and is associated with significant burden. Highly effective treatments exist for PTSD, evidence-based psychotherapies, but very few Veterans receive them. Although VA has trained over 8,500 providers in evidence-based psychotherapies for PTSD over the past 10 years, only 6% of the 650,000 VHA patients with PTSD receive an evidence-based psychotherapy. It is critical to connect Veterans with the most effective PTSD treatments and done so in a way that is Veteran-centered. Shared decision making is a patient-centered approach to choosing healthcare treatment options. It has been shown to increase patients' motivation for treatment and ability to stay in treatment long enough to get benefit. It has also been shown to help providers align their practice with evidence-based guidelines. This proposal will refine and pilot test a shared decision making intervention for PTSD to be used in VA primary care clinics, where the vast majority of Veterans with PTSD are treated.

DETAILED DESCRIPTION:
Background: Over 1 million Veterans have PTSD and most (80% or more) do not receive first-line treatments, evidence-based psychotherapies, despite significant VA investment to increase access to these treatments. Clinicians often struggle to engage Veterans in evidence-based psychotherapies because they can be emotionally challenging treatments. Engagement could be catalyzed by mental health providers integrated into primary care (i.e., VA's Primary Care-Mental Health Integration, or PC-MHI) to maximize the reach of engagement efforts beyond specialty PTSD settings. Shared decision making, a process by which the patient and provider discuss treatment options, weigh benefits and risks, and select a treatment that meets the patient's needs, addresses known patient and provider barriers to evidence-based psychotherapies, including knowledge, self-efficacy, and trust. However, no study has examined shared decision making for PTSD in primary care. The proposal will address this knowledge gap by developing and refining a shared decision making intervention for PTSD, Patient Readiness for Improvement through Motivation, Engagement, and Decision-making (PRIMED), using input from Veterans with diverse perspectives, PC-MHI providers, and VA operational partners to optimize integration of shared decision making into clinical care. The investigators will collect acceptability and feasibility data to support an application for a future effectiveness-implementation trial.

Significance/Impact: Dr. Chen's proposed research addresses three HSR&D and VA priorities: 1) increase engagement and retention of Veterans in evidence-based PTSD treatments, 2) advance health services research methods, specifically implementation science and user-centered design, which focuses on thorough integration of Veteran and frontline provider input, and 3) support suicide prevention efforts through effective treatment of PTSD, a major risk factor for suicide.

Innovation: The proposed project will promote significant change in current VA clinical practice. PC-MHI providers typically refer out patients with PTSD and defer discussions about treatment options to specialty providers. This proposal will help PC-MHI providers use a formal engagement strategy, shared decision making, to improve patients' knowledge of first-line PTSD treatments and to build motivation for care.

Specific Aims: 1) Refine PRIMED using user-centered design methods and diverse Veterans' perspectives, 2) Beta test PRIMED in one rural and one urban PC-MHI clinic to optimize integration into clinical workflow and achieve satisfactory acceptability and feasibility across a range of settings, 3) Conduct a small, randomized pilot trial (N=40) of PRIMED vs. usual care in two VA PC-MHI clinics to assess the feasibility of study procedures, which will inform a future larger trial.

Methodology: In Aim 1, Dr. Chen will conduct qualitative interviews using user-centered design methods with 25 VA PC-MHI patients with PTSD, oversampling women veterans and racial/ethnic minority veterans, to refine the PRIMED intervention protocol. In Aim 2, Dr. Chen will use rapid, iterative beta-testing with approximately 20 patients to optimize the acceptability and feasibility of delivering PRIMED in the clinical setting and its integration into clinical workflow across varied settings (small rural clinics and large urban clinics). In Aim 3, Dr. Chen will conduct a pilot randomized feasibility trial (N=40) to assess the feasibility of recruiting and randomizing Veterans and measuring treatment engagement and clinical outcomes.

Next Steps/Implementation: The research and training activities will prepare the nominee to conduct a multi-site, hybrid type 1 effectiveness-implementation trial to test the effectiveness of PRIMED for increasing receipt of first-line PTSD treatments and to begin to assess implementation barriers and facilitators. Future work to move this research into practice would involve collaborating with operational partners to improve VA SAIL performance measures in mental health, which are weighted to encourage evidence-based psychotherapies.

ELIGIBILITY:
Inclusion Criteria:

* Adult VA patients 18 years who have a documented initial visit to Primary Care-Mental Health Integration for PTSD in the past 90 days at VA Puget Sound

Exclusion Criteria:

* Cognitive impairment (e.g., moderate or severe history of traumatic brain injury, dementia)
* Unstable acute psychiatric conditions (e.g., current high-risk for suicide)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
CollaboRATE | 2 weeks
  CollaboRATE is a a 3-item instrument developed for measuring patient-centeredness within SDM. Good patient acceptability will be defined as minimum ratings of 3 (some effort was made) on a 0 (no effort was made) to 4 (every effort was made) scale for every one of the 3 questionnaire items: 1) How much effort was made to help you understand your health issues?, 2) How much effort was made to listen to the things that matter most to you about your health issues?, 3) How much effort was made to include what matters most to you in choosing what to do next?
Utilization of evidence-based psychotherapies (EBPs) for PTSD | 6 months
  The investigators will use chart review methods to identify utilization of EBPs. One method is as a dichotomous (yes/no) measure of initiation.
Utilization of evidence-based psychotherapies (EBPs) for PTSD | 6 months
  The investigators will measure the number of EBP sessions received in 6 months.
Utilization of evidence-based psychotherapies (EBPs) for PTSD | 6 months
  The investigators will measure time to initiation, defined as days between the initial PC-MHI triage visit and first EBP session.

SECONDARY OUTCOMES:
PTSD Knowledge Questionnaire | 2 weeks
  Knowledge about PTSD and its treatment will be assessed with a 43-item true-or-false questionnaire, which was used in a previous RCT of a paper-based PTSD decision aid. Items will rated as o (incorrect) or 1 (correct), with a total score ranging from 0-43. Higher scores indicate more accurate knowledge.
Decisional Conflict Scale | 2 weeks
  The DCS is a 16-item scale that assesses patient-reported uncertainty around treatment decision-making. The items also assess the degree to which patients feel informed about risks and benefits, clear about their personal attitudes and values, supported by other(s), and effective in decision making. The items are rated from 0 (strongly agree) to 4 (strongly disagree), with a range from 0 to 64. Higher scores indicate better outcomes, i.e., more confidence and feeling more informed.
Perceived Stigma and Barriers to Care for Psychological Problems | 2 weeks
  The investigators will use a 10-item version adapted for Veterans to assesses perceived barriers to mental health treatment related to access, stigma, and trust in providers. Higher scores indicate worse outcomes, i.e., more perceived stigma and barriers to care.
Generalized Self-Efficacy | 2 weeks
  A 10-item scale that measures an individual's perceived ability to problem solve, follow through with decisions, and cope effectively with challenges. Items are rated from 0 (not at all true) to 4 (exactly true) and summed. Higher scores indicate better outcomes, i.e., greater confidence.
Wake Forest Physician Trust Scale | 2 weeks
  A 10-item scale that measures patients' trust in their care providers. The scale total ranges from 10 to 50. Higher scores indicate more trust. Example questions include "Sometimes your doctor cares more about what is convenient for [him or her] than about your medical needs" and "Your doctor is totally honest in telling you about all of the different treatment options available for your condition." The language will be adapted so that "mental health provider" replaces "doctor" to clearly indicate to patients the relationship of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica A. Chen, PhD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No